CLINICAL TRIAL: NCT03827733
Title: Gut Microbiota and Alzheimer's Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Yuan Shen, MD, PhD, Chief of Psychiatry Department, Shanghai 10th People's Hospital
Other Study IDs: dsyy004
Record Dates: First submitted 2018-11-28; First posted 2019-02-01 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer Disease
Keywords: Gut Microbiota; Alzheimer's Diseases
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fecal sample collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AD patients: Participants who are diagnosed with AD.
- Partners of the AD patients: Partners of AD patients who live together with the AD patients.
- Elderly participants with normal cognition: Community dwelling elderly with normal cognition and with AD.

SUMMARY:
The investigator will perform clinical studies to test a hypothesis that participants who have Alzheimer's disease will have different gut/oral microbiota profile as compared to the participants who do not have Alzheimer's disease. The investigators will also check the microbiome of their partners in this study. The investigators plan to perform the studies in 150 participants in Shanghai Tenth's People's Hospital and also in the houses in Shanghai city. Investigators will also measure the beta-amyloid in the feces of the participants. Finally, the investigators will determine cognitive function in these participants.

DETAILED DESCRIPTION:
Studies have shown that gut/oral microbiome and beta-amyloid in body may have a significant impact on the behavior and brain pathology consistent with Alzheimer's disease (AD) neuropathogenesis. The objective of this study is to assess whether the gut/oral microbiome and feces beta-amyloid of AD patients are different from those of the participants without AD and their partners. The investigators plan to recruit 150 subjects, including three groups of normal elders, AD patients and the partners of the AD patients. The cognitive function will be assessed and the feces and oral samples will be collected to determine whether there are differences or correlations.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 and older

Exclusion Criteria:

* with other acute gastrointestinal diseases
* with other severe neuropsychiatric disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly participants with normal congition will be collected from community. Alzheimer's disease participants and their spouse will be collected from Shanghai Tenth People's Hopital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut beta-amyloid 42 | Through study completion, an average of 4 year
  Gut amyloid-beta 42 will be determined by digital ELISA, traditional ELISA and western blot.

SECONDARY OUTCOMES:
Gut microbiota | Through study completion, an average of 4 year
  We will use DNA sequencing to define the profile of gut microbiota.
Oral microbiota | Through study completion, an average of 4 year
  We will use DNA sequencing to define the profile of gut microbiota.
Cognitive function by Mini-mental State Examination (MMSE) | through study completion, an average of 4 year
  We will assess the cognitive function in the participants using MMSE to promote the diagnosis of AD in these participants. The sum of MMSE ranges from 0 (worse) to 30 (better).

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shen, MD, PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided